CLINICAL TRIAL: NCT06703905
Title: Short and Long-term Outcomes of Minimally Invasive Pancreatoduodenectomy Combined with Triangle Operation for Resectable Pancreatic Cancer: an International Multicenter Randomized Controlled Study
Brief Title: Conventional Partial Pancreatoduodenectomy Versus an Extended Pancreatoduodenectomy for Pancreatic Head Cancers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZXIIT2024180
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Cancer Resectable
Keywords: Pancreatic cancer; pancreaticoduodenectomy; Minimally invasive surgery; Heidelberg Triangle
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PD group (Active Comparator): Traditional minimally invasive pancreaticoduodenectomy
  Interventions: Procedure: Pancreaticoduodenectomy
- expanded PD group (Experimental): Traditional minimally invasive pancreaticoduodenectomy combined with the TRIANGLE procedure
  Interventions: Procedure: Expanded pancreaticoduodenectomy surgery

INTERVENTIONS:
Procedure: Expanded pancreaticoduodenectomy surgery — Traditional minimally invasive pancreaticoduodenectomy combined with the TRIANGLE procedure
  Arms: expanded PD group
Procedure: Pancreaticoduodenectomy — Traditional minimally invasive pancreaticoduodenectomy
  Arms: PD group

SUMMARY:
The goal of this clinical trial is to learn if traditional pancreaticoduodenectomy (PD) combined with TRIANGLE (extended PD surgery) can increase disease-free survival (DFS) in patients with pancreatic head cancers compared to traditional minimally invasive PD. The main questions it aims to answer are:

* Does extended PD surgery increase disease-free survival (DFS)?
* Does extended PD surgery could improve postoperative and long-term quality of life for patients? Researchers will compare extended PD surgery to traditional PD surgery to see if extended PD surgery could extend the survival time of patients.

Participants will:

* Accept traditional minimally invasive PD surgery or minimally invasive PD combined with TRIANGLE surgery.
* Visit the clinic once every 3 months for checkups and tests.
* Keep a diary of their symptoms.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) currently stands as the sole option for treating resectable pancreatic head cancer; however, the long-term post-operative survival quality of patients remains unpromising. According to statistics from international multicenter studies, the 5-year survival rate of patients post-surgery does not exceed 20%. The principal causes for the suboptimal survival quality are the high recurrence and metastasis tendencies of pancreatic cancer, along with its low sensitivity and poor response to the existing neoadjuvant therapy. In contrast to traditional PD, PD combined with the TRIANGLE procedure (expanded PD) enables more thorough resection, effectively addressing the early recurrence and metastasis issues of pancreatic cancer and holds significant potential in enhancing patients' long-term survival quality. Nevertheless, there exists no high-level clinical evidence regarding the improvement of short-term complications for this surgical approach. Simultaneously, minimally invasive pancreatic surgeries have been demonstrated in high-throughput pancreatic centers to improve patients' short-term quality of life, yet the effect on long-term prognosis remains ambiguous. Hence, our center innovatively proposes minimally invasive PD in combination with the TRIANGLE procedure for the treatment of resectable pancreatic cancer, with the aim of integrating the advantages of both intervention measures to improve patients' post-operative quality of life and long-term survival quality.

This research will carry out a randomized controlled trial on patients with resectable pancreatic cancer who are scheduled to undergo minimally invasive PD in six Chinese centers and two foreign centers, comparing the prognostic disparities between traditional PD and the expanded PD procedure. The primary outcome measure is the postoperative disease-free survival (DFS), defined as "the time from randomization to disease recurrence or death for any reason." The projected enrollment period is 15 months, and the follow-up duration is 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative: a. Patients with suspected or histologically verified resectable, borderline or locally advanced pancreatic cancer of the pancreatic head (i.e. pancreatic ductal adenocarcinoma, intraductal papillary mucinous neoplasm (IPMN)-carcinoma or periampullary cancer of the pancreatobiliary-type) ; b. Patients scheduled for elective partial pancreatoduodenectomy (irrespective of neoadjuvant therapy); c. Assumed resectability in accordance with the surgical protocol for experimental and control intervention as judged by the treating surgeon; d. Ability of the subject to understand character and individual consequences of the clinical trial;e.Written informed consent; f. Age ≥ 18 years;
2. Intraoperative: a.No distant metastases; b.No paraaortic lymph node metastases; c.Intraoperative confirmation that the patient can be operated on according to both surgical methods.

Exclusion Criteria:

1. Participation in another interventional trial with the interference of intervention and outcome of this trial;
2. American Society of Anesthesiologists (ASA) grade >3;
3. Distant metastatic disease .

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 270 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival after resection | 3, 6, 12, 18, 24, 30, 36 months after surgery (or early termination of the trial)
  the primary outcome was DFS defined "as the time from randomisation until disease recurrence or death from any cause"

SECONDARY OUTCOMES:
the rate of microscopically complete margin clearance | Intraoperative
  the rate of >0.1 cm margin clearance, R0(CRM-)
the rate of microscopic margin clearance ≤ 0.1 cm | Intraoperative
  rate of R0(CRM+)
the rate of microscopic margin involvement (R1) resections | Intraoperative
  the rate of R1 resection, defined according to the 8th edition of the UICC TNM classification
the rate of postoperative pancreatic fistula | Day of discharge, postoperative days 5, 10-12 and 90
  the POPF was defined by the International Study Group of Pancreatic Surgery (ISGPS)
the rate of postpancreatectomy haemorrhage | Day of discharge, postoperative days 5, 10-12 and 90
  PPH was defined by the ISGPS
the rate of delayed gastric emptying | Day of discharge, postoperative days 5, 10-12 and 90
  DGE was defined by the ISGPS
the rate of bile leakage | Day of discharge, postoperative days 5, 10-12 and 90
  Bile leakage was defined by the International Study Group of Liver Surgery (ISGLS)
the rate of lymphatic fistula | Day of discharge, postoperative days 5, 10-12 and 90
  Lymphatic fistula was defined by the ISGPS
the rate of diarrhoea | Day of discharge, postoperative days 5, 10-12 and 90
  Diarrhoea was graded by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

OTHER OUTCOMES:
Overall survival | 3, 6, 12, 18, 24, 30, 36 months after surgery (or early termination of the trial)
Quality of Life questionnaire (QLQ-C30) | Screening, Day of discharge, and 6, 12, 18, 24, 30, 36 months after surgery
  Defined according to the European Organisation for Research and Treatment of Cancer (EORTC) Core Quality of Life questionnaire QLQ-C30
pancreatic cancer specific questionnaire (PAN26) | Screening, Day of discharge, and 6, 12, 18, 24, 30, 36 months after surgery
  The European Organisation for Research and Treatment of Cancer (EORTC) pancreatic cancer specific questionnaire (QLQ-PAN26)
Local recurrence within the study period | 3, 6, 12, 18, 24, 30, 36 months after surgery (or early termination of the trial)
Length of primary hospital stay in days | Day of discharge
  Length of primary hospital stay in days was from the day of index operation to the day of discharge
Quality of recovery | Screening, postoperative days 5
  Defined according to the QoR-15 questionnaire on postoperative day 5 compared to baseline
Serious adverse events | Day of surgery, day of discharge, postoperative days 5, 10-12 and 90, and 6, 12, 18, 24, 30, 36 months after surgery (or early termination of the trial)

IPD SHARING:
Plan to Share IPD: Undecided